CLINICAL TRIAL: NCT01502384
Title: A Longitudinal Study in 1st Degree Relatives of Parkinson's Disease (PD) Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Beth Israel Medical Center (Other); Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: TASMC-11-NG-0463
Record Dates: First submitted 2011-12-28; First posted 2011-12-30 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Parkinson's Disease
Keywords: healthy 1st degree relatives of pd patients
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy relatives: healthy 1st degree relatives of PD patients
  Interventions: Other: neurological examination

INTERVENTIONS:
Other: neurological examination — motor and cognitive functions

SUMMARY:
This is a longitudinal study in healthy 1st degree relatives of patients with Parkinson's Disease (PD) carriers of a genetic mutation in genes that are known to increase the risk for PD. The purpose of this study is to explore the association between genetic mutations in the known genes and early preclinical symptoms such as motor, sensory, autonomic, behavioral and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* healthy 1ST degree relatives of PD patients with known genotype that participated in an earlier genetic study at the sourasky medical center.

Exclusion Criteria:

* subjects with cognitive decline by the parameters defined in DSM- IV
* subjects with psychiatric disorder
* subjects unable to sign a consent form

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy 1ST degree realtives of PD patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Di Monte DA. The environment and Parkinson's disease: is the nigrostriatal system preferentially targeted by neurotoxins? Lancet Neurol. 2003 Sep;2(9):531-8. doi: 10.1016/s1474-4422(03)00501-5. PMID 12941575
- [Background] Di Monte DA, Lavasani M, Manning-Bog AB. Environmental factors in Parkinson's disease. Neurotoxicology. 2002 Oct;23(4-5):487-502. doi: 10.1016/s0161-813x(02)00099-2. PMID 12428721
- [Background] Huang Y, Cheung L, Rowe D, Halliday G. Genetic contributions to Parkinson's disease. Brain Res Brain Res Rev. 2004 Aug;46(1):44-70. doi: 10.1016/j.brainresrev.2004.04.007. PMID 15297154
- [Background] Quik M. Smoking, nicotine and Parkinson's disease. Trends Neurosci. 2004 Sep;27(9):561-8. doi: 10.1016/j.tins.2004.06.008. PMID 15331239
- [Background] Vila M, Przedborski S. Genetic clues to the pathogenesis of Parkinson's disease. Nat Med. 2004 Jul;10 Suppl:S58-62. doi: 10.1038/nm1068. PMID 15272270
- [Background] von Bohlen und Halbach O, Schober A, Krieglstein K. Genes, proteins, and neurotoxins involved in Parkinson's disease. Prog Neurobiol. 2004 Jun;73(3):151-77. doi: 10.1016/j.pneurobio.2004.05.002. PMID 15236834
- [Background] Farrer M, Stone J, Mata IF, Lincoln S, Kachergus J, Hulihan M, Strain KJ, Maraganore DM. LRRK2 mutations in Parkinson disease. Neurology. 2005 Sep 13;65(5):738-40. doi: 10.1212/01.wnl.0000169023.51764.b0. PMID 16157908
- [Background] Wilk JB, Lash TL. Risk factor studies of age-at-onset in a sample ascertained for Parkinson disease affected sibling pairs: a cautionary tale. Emerg Themes Epidemiol. 2007 Apr 4;4:1. doi: 10.1186/1742-7622-4-1. PMID 17408493
- [Background] Orr-Urtreger A, Shifrin C, Rozovski U, Rosner S, Bercovich D, Gurevich T, Yagev-More H, Bar-Shira A, Giladi N. The LRRK2 G2019S mutation in Ashkenazi Jews with Parkinson disease: is there a gender effect? Neurology. 2007 Oct 16;69(16):1595-602. doi: 10.1212/01.wnl.0000277637.33328.d8. PMID 17938369
- [Background] Clark LN, Nicolai A, Afridi S, Harris J, Mejia-Santana H, Strug L, Cote LJ, Louis ED, Andrews H, Waters C, Ford B, Frucht S, Fahn S, Mayeux R, Ottman R, Marder K. Pilot association study of the beta-glucocerebrosidase N370S allele and Parkinson's disease in subjects of Jewish ethnicity. Mov Disord. 2005 Jan;20(1):100-3. doi: 10.1002/mds.20320. PMID 15517591
- [Background] Thaler A, Ash E, Gan-Or Z, Orr-Urtreger A, Giladi N. The LRRK2 G2019S mutation as the cause of Parkinson's disease in Ashkenazi Jews. J Neural Transm (Vienna). 2009 Nov;116(11):1473-82. doi: 10.1007/s00702-009-0303-0. PMID 19756366
- [Background] Mirelman A, Gurevich T, Giladi N, Bar-Shira A, Orr-Urtreger A, Hausdorff JM. Gait alterations in healthy carriers of the LRRK2 G2019S mutation. Ann Neurol. 2011 Jan;69(1):193-7. doi: 10.1002/ana.22165. PMID 21280089